CLINICAL TRIAL: NCT04544982
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy of Blue Fenugreek Kale Extract (BFKE) on Skin.
Brief Title: Study to Evaluate the Efficacy of Blue Fenugreek Kale Extract (BFKE) on Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MGB/191101/BFKE/SKNM
Record Dates: First submitted 2020-08-26; First posted 2020-09-10 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2020-09

CONDITIONS: Skin Health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue fenugreek kale extract (Active Comparator): One capsule to be taken orally before breakfast and one capsule after lunch, with water.
  Interventions: Other: Blue fenugreek kale extract
- Placebo (Placebo Comparator): One capsule to be taken orally before breakfast and one capsule after lunch, with water.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Blue fenugreek kale extract — One capsule to be taken orally before breakfast and one capsule after lunch, with water.
  Arms: Blue fenugreek kale extract
Other: Placebo — One capsule to be taken orally before breakfast and one capsule after lunch, with water.
  Arms: Placebo

SUMMARY:
Participants will be supplemented BFKE for a period of 8-weeks to improve skin health. The objective of the study is to evaluate the 'Transepidermal Water Loss (TEWL)' that characterizes the skin barrier function of stratum corneum. Additional parameters include, evaluation of skin moisture content, wrinkling, elasticity, sagging, radiance and also on inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult female participants aged ≥ 30 and ≤ 55 years.
* Participants with signs of poor skin barrier as determined by Trans-epidermal water loss ≥ 15 g/m2/h on forehead.
* Participants with skin type II to IV as per Fitzpatrick skin type calculator.
* Participants with skin type II and III as per Glogau's classification of photoageing skin.
* Participants must have Body Mass Index (BMI) ≥ 18.5 ≤ 29.9 kg/m2.
* Participants with moderate signs of Melasma as assessed by the investigators.
* Participants ready to abstain from any cosmetic or drug-based cream, ointment, lotion and other products apart from the ones allowed during study period.
* Participants ready to rinse their face only with water and to refrain from using soap, facewash, make-up etc. or any other cosmetic care related products 12 hrs. prior to any assessment visit.

Exclusion Criteria:

* Unwilling to forgo any aesthetic or dermatological treatments or procedures during the study period.
* Participants with visible scarring on face.
* Participants having any form of skin disorder on the Nasolabial fold.
* Water consumption history of ≤ 500 ml and ≥ 3000 ml per day.
* Smoking or using any tobacco products.
* Participants presently undergoing or had undergone treatment for softening or reducing wrinkles in the last 3 months.
* Having a history of chronic skin allergies.
* History of heavy caffeine usage ≥ 4 cups in a day.
* Binge drinkers as defined by consumption of 4 or more alcohol containing beverages within 2 hours.
* Presence of unstable, acutely symptomatic, or life-limiting illness.
* Participants taking any vitamins and other related supplements.
* Menopausal and peri-menopausal females.
* Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
* Females who have had participated in a study of an investigational product 90 days prior to the screening.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Trans Epidermal Water Loss (TEWL) using Tewameter®. | From Base line Day 0 to day 56
  To evaluate the effect of 8-week consumption of BFKE on skin barrier function as evaluated by Trans Epidermal Water Loss (TEWL) using Tewameter®.
Skin moisture | From Base line Day 0 to day 56
  skin hydration as measured by skin moisture (forehead & forearm) using skin moisture analyzer.
Modified Fitzpatrick Wrinkle Severity Scale | From Base line Day 0 to day 56
  Changes in the wrinkle class from Class 3.0 indicated worst means Deep wrinkle. Deep and furrow wrinkle; more than 3-mm wrinkle depth to Class 0 indicates Good means No wrinkle. No visible wrinkle; continuous skin line.
Ezure Sagging scale | From Base line Day 0 to day 56
  Cheek with Highest sagging score means Very severe sagging indicates worst and Lowest sagging score means No sagging indicates better
Pinch recoil test | From Base line Day 0 to day 56
  A decrease in pinch recoil time is associated with improvement in skin elasticity/firmness.
Skin parameters using a participant based self-assessment questionnaire | From Base line Day 0 to day 56
  Highest Score represents Better and lowest Score represents Worst
Investigator's global assessment using 5-point Likert scale | From Base line Day 0 to day 56
  The Study Investigator will assess on a scale of 0 (Very poor) to 4 (Excellent) as to how beneficial or vice-versa was the treatment experience over the study period.
Participant's global assessment using 5-point Likert scale | From Base line Day 0 to day 56
  The Participant will self-assess on a scale of 0 (Very poor) to 4 (Excellent) as to how beneficial or vice-versa was the treatment experience over the study period.
Inflammatory biomarkers | From Base line Day 0 to day 56
  Change in the levels of Inflammatory biomarkers within specified range
Allergic skin inflammation as assessed by Eosinophil to basophil ratio and Neutrophil to lymphocyte ratio. | From Base line Day 0 to day 56
  Change in the levels of Eosinophil to basophil ratio and Neutrophil to lymphocyte ratio within specified range
Oxidative Stress as assessed by Malondialdehyde concentration. | From Base line Day 0 to day 56
  malondialdehyde concentration of the samples will be measured as an index of lipid peroxidation

CONTACTS AND LOCATIONS:
Locations (1):
- Skin cure and care clinic, Thane, Maharashtra, India